CLINICAL TRIAL: NCT05364632
Title: Effects of Aerobic Training Versus Behavioral Intervention to Increase Physical Activity in Patients With Asthma: a Randomized, Blinded Clinical Trial.
Brief Title: Aerobic Training Versus Behavioral Intervention to Increase Physical Activity in Patients With Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Celso R. Carvalho, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/03745-3
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Asthma
Keywords: asthma; physical activity; physical exercise; quality of life
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Evaluations will be conducted blindly, that is, by an evaluator who will not be directly involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Intervention (Experimental): Participants will undergo an eight-week behavioral intervention protocol (once a week) aimed at increasing the level of physical activity, consisting of a brief educational program: brief education for asthma and benefits of physical activity and behavioral intervention based on Social Cognitive Theory and the Theory of Stages of Behavior Change.
  Interventions: Behavioral: Behavioral Intervention to Increase Physical Activity
- Aerobic Training (Experimental): Participants will undergo an eight-week aerobic training protocol (twice a week) on a treadmill, each aerobic training session will consist of 45 minutes divided into 5 minutes of warm-up, 35 minutes of aerobic exercise and 5 minutes of cool-down.
  Interventions: Other: Aerobic Training

INTERVENTIONS:
Behavioral: Behavioral Intervention to Increase Physical Activity — The educational program will consist of 2 classes held once a week, each lasting 90 minutes. The classes will be based on an education videotape, presentations and group discussions. The first class will address the asthma education. The second class will be about the current international physical activity recommendations and the importance and benefits of being physically active. The behavioural intervention will be performed in 8 weekly goal-setting consultation, face-to-face, each lasting until 90 minutes. Patients will be offered a commercially-available activity tracker to wear during 3 days prior to each consultation. According to their own physical activity (PA) data and the behavioural change stage, an individual action plan will be established to increase physical activity. Each participant will receive individual counselling with the goal of increasing participation in PA and reducing their sedentary time.
  Arms: Behavioral Intervention
Other: Aerobic Training — The same initial educational program described for the Behavioral Intervention group will be delivered to this group. Each aerobic training session will consist of 45 minutes divided into 5 minutes of warm-up, 35 minutes of aerobic exercise and 5 minutes of cool-down. During physical training, heart rate and level of respiratory distress will be monitored. The intensity of aerobic physical training will be based on the heart rate (HR) corresponding to one third of the difference between the anaerobic threshold (LA) and the respiratory compensation point (CRP). The patient may interrupt physical exercise if he presents any clinical symptoms and/or respiratory discomfort, returning as soon as his respiratory condition improves.
  Arms: Aerobic Training

SUMMARY:
To compare the effects of aerobic training and behavioural intervention to increase physical activity in the clinical control of asthma and in the quality of life of patients with asthma.

DETAILED DESCRIPTION:
Adult participants of both genders with moderate to severe asthma, not physically active, will be evaluated after being informed about the study, agreeing and signing the informed consent form. Participants will be randomized to aerobic training or behavioral intervention group. Both interventions will consist of 8 weeks. Aerobic training will be performed on a treadmill (2xweek; 45 min/session). The behavioral intervention will be a program to increase physical activity (1xweek; up to 90 min / session). The maximum HR will be estimated according to the Tanaka's equation (208 - 0.7 x age).

ELIGIBILITY:
Inclusion Criteria:

1. Participants not physically active;
2. Uncontrolled asthma (ACQ>1,5);
3. Diagnosis of asthma based on the recommendations of the Global Initiative for Asthma (GINA 2020);
4. Be under outpatient follow-up at the Pulmonology or Immunology service of the University of Sao Paulo General Hospital;
5. Be under outpatient medical treatment for at least six months, with a stable clinical condition for at least 30 days;
6. Being using optimized drug therapy for asthma.

Exclusion Criteria:

1. Participation in another research protocol;
2. Difficulty in understanding any of the questionnaires used;
3. Practitioners of regular physical activity;
4. Pregnancy and psychiatric problems that make it difficult to understand the questionnaires and the study protocol;
5. Presence of another chronic lung, neurological or musculoskeletal disease that hinders or prevents physical activity;
6. Patients who are smokers or ex-smokers (who have quit smoking for less than 1 year or who have smoked more than 15 pack-years).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in asthma clinical control | [Change from baseline at 8 weeks of intervention and at 16 weeks post intervention]
  Clinical control will be evaluated by the Asthma Control Questionnaire (ACQ). The ACQ contains 7 items rated on a 7- point scale (0 = without limitation, 6 = maximum limitation), with a higher score indicating worse control. Scores lower than 0.75 are associated with good asthma control, whereas scores greater than 1.5 are indicative of poorly controlled asthma, and a change of at least 0.5 points in the ACQ score is regarded as clinically significant.

SECONDARY OUTCOMES:
Change in sedentary behaviour | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Sedentary behaviour will be objectively quantified using a movement sensor (ActiGraph, Pensacola, USA) for 7 consecutive days on the hip using an elastic belt. Sedentary behaviour will be quantify by the time spent sedentary (<100 counts/min).
Change in physical activity levels | [Time Frame: Change from baseline at 8 weeks of intervention and at 16 weeks post intervention]
  Physical activity will be objectively quantified using a movement sensor (ActiGraph, Pensacola, USA) for 7 consecutive days on the hip using an elastic belt.
Change in Health Factors Related to Quality of Life in Asthma | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Health related quality of life will be assessed by Asthma Quality Life Questionnaire (AQLQ). The AQLQ consists of 32 items rated on a 7-point scale (1 = great deal, 7 = not at all) divided into the following 4 domains: activity limitations, symptoms, emotional function and environmental stimuli. Higher AQLQ scores indicate a better quality of life, and treatments resulting in a 0.5-point increase in scores following an intervention are considered to be clinically effective.
Change in psychosocial symptoms | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Symptoms of anxiety and depression symptoms will be assessed by the Hospital Anxiety and Depression scale (HADs), which consists of 14 items divided into 2 subscales (7 for anxiety and 7 for depression). Each item is scored from 0 to 3, with a maximum score of 21 points for each subscale. A score greater than 8/9 in each subscale suggests a diagnosis of either anxiety and/or depression.
Change in body composition - Weight | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Bioimpedance (Octopolar InBody 720).
Change in body composition - Fat mass | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Bioimpedance (Octopolar InBody 720).
Change in body composition - Visceral adiposity area | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention.
  Bioimpedance (Octopolar InBody 720). ,Fat-free mass, and skeletal muscle mass will be calculated.
Change in body composition - Fat-free mass | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention]
  Bioimpedance (Octopolar InBody 720).
Change in body composition - Skeletal muscle mass | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention]
  muscle mass Bioimpedance (Octopolar InBody 720).

OTHER OUTCOMES:
Changes in Barriers to the practice of Physical Activities of Daily Living | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention]
  The possible answers to the questionnaire Barriers to the practice of Physical Activities of Daily Living are never, rarely, sometimes, almost always or always and the score for each item varies from 0 to 4. It will be considered as limiting domain for physical activities those in which individuals report a value equal to or greater than 3 in at least half of the barriers.
Change in asthma exacerbation | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Asthma exacerbation will be assessed by the following criteria: the use of ≥4 puffs of rescue medication per 24 hours during a 48-hour period, a need for systemic corticosteroids, an unscheduled medical appointment, and either a visit to an emergency room or hospitalization
Change in Behavioral Stage for physical activity practice | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  The Behavioral Stage Assessment Questionnaire for the Practice of Physical Activity qualitatively assesses thinking in relation to the practice of physical activity, and may present the following stages of behavior: 1. Pre-contemplation; 2.
  Contemplation; 3. Preparation; 4. Action; 5- Maintenance.
Pulmonary function | Baseline
  Lung volumes will be assessed by spirometry
Change in anthropometric indexes | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  Waist circumference (cm) and hip circumference (cm) will be combined to report wait to hip ratio (WHR).
Sleep quality assessment | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  The assessment of sleep quality will be performed by the accelerometer (Actigraph, GT9) for seven nights before and after the interventions, throughout the day. The outcomes derived from the monitor will be sleep latency (the amount of time needed to fall asleep) and sleep efficiency (number of sleep minutes divided by the total number of minutes the participant was in bed).
Cardiopulmonary Exercise Test | Change from baseline at 8 weeks of intervention and at 16 weeks post intervention
  CPET will be performed on an electric cycle ergometer (Corival; Lode BV Medical Technology, Netherlands) equipped with an electronic system (CPX System; CareFusion, Germany). During the test there will be verbal encouragement for the patient to reach maximum effort. The maximum oxygen consumption (VO2 peak in ml.kg.min) will be evaluated, considered the highest value in the test phase; anaerobic threshold (will be determined from the exponential growth of ventilation, additionally by the increase in VCO2, fall and/or stabilization of VO2, also considering the VCO2/VO2 ratio close to 1; respiratory compensation point (will be determined from the second point inflection, exponential growth in ventilation, additionally due to the increase in VCO2 and exponential fall in VO2, also considering the VCO2/VO2 ratio greater than or equal to 1.10; maximum heart rate (established by electrocardiogram examinatio).

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Clinical Hospital of São Paulo University medical school (HCFMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Araujo Pinheiro DH, Silva RAD, Lunardi AC, Cervera VZ, Carvalho-Pinto RM, de Lima FF, Carvalho CRF. Effects of Aerobic Training Versus Behavioral Intervention to Increase Physical Activity for Disease Control in Patients With Asthma: Protocol for a Randomized Trial. JMIR Res Protoc. 2025 Oct 30;14:e78603. doi: 10.2196/78603. PMID 41166708